CLINICAL TRIAL: NCT01129505
Title: Preventing Childhood Obesity: Early Intervention During Pregnancy and First Year Postpartum for Overweight and Obese Women Using a Two-pronged Family-based Nutrition & Exercise Lifestyle Intervention Program (NELIP).
Brief Title: Preventing Childhood Obesity: A Two-pronged Approach Starting in Pregnancy and the First Year Postpartum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Health Research Foundation (Other)
Responsible Party: Principal Investigator, Michelle Mottola, Dr. Michelle F. Mottola, FACSM, University of Western Ontario, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OPG-92367
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Childhood Obesity; Excessive Weight Gain in Pregnancy With Baby Delivered; Dietary Modification; Healthy Lifestyle Habits
Keywords: pregnancy; intervention; exercise; nutrition; infants
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Nutrition & Exercise Lifestyle Intervention Program (NELIP) — Nutrition- individualize total energy intake with a minimum of 2000 kcal/day with a restriction of not more than 33% total energy intake, total carbohydrate of 40-50% total energy intake, total fat intake of 30% of total energy intake (substituting monounsaturated fatty acids for saturated and trans-fatty acids), and approximately 30% dedicated to protein intake.
  Exercise-25 minutes of walking per session, 3-4 times per week, each subsequent week increasing by 2 mins to a maximum of 40 mins/session.
  Family-based Behavioural Treatment (FBBT) Coupled with the individualized NELIP for each woman, FBBT will be presented in 3 group sessions (including family members), focussing on strategies to make healthy lifestyle choices with behavioural strategies.
  Other Names: NELIP; FBBT

SUMMARY:
Our longitudinal aim is to reduce childhood obesity using our two-pronged intervention program, which includes healthy food choices and increased physical activity initiated during pregnancy and re-instated in the early period after delivery for overweight and obese women. We will accomplish this with our family-based Nutrition and Exercise Lifestyle Intervention Program (NELIP) to promote healthy family living. An intervention targeting school-aged children on the importance of healthy lifestyles occurs too late to prevent childhood obesity and establish lifelong healthy body weights. To break this spiraling cycle of generations of unhealthy body weights in Canadian children, and to reduce the risk of future obesity-related health problems, it is necessary to prevent excessive pregnancy weight gain, high blood sugars in the mother and to promote a healthy lifestyle during pregnancy and early post delivery. With our NELIP team as a cornerstone, and our pilot data already collected with promising results, we foresee an opportunity over the next 3 years to contribute to changing patient care with emphasis on disease prevention and healthy family lifestyle initiation early in life to reverse the trend of childhood obesity. With a solid research-based initiative from the lab to the community by educating health care providers, future health care can be improved by putting prevention-based programs into practice.

Healthy women = healthy babies = healthy families = healthy futures!!

DETAILED DESCRIPTION:
Overweight and obesity have been identified as major neglected public health issues, as the prevalence of unhealthy body weights is increasing world-wide at an alarming rate. There is a robust link between the fetal environment and its long-term influence on health and susceptibility to future chronic disease in the offspring. Obesity begets obesity, and an unhealthy maternal metabolic state can have a profound influence on the risk of early obesity development in the child. Excessive pregnancy weight gain and high pre-pregnant body-mass index (BMI) have been linked to gestational diabetes (GDM) and macrosomic infants (birth weight >4.0kg. Since much of the influence of the intrauterine milieu is transmitted to the next generation non-genetically, potentially deleterious effects can be reversed and prevented. An intervention targeting school-aged children on the importance of healthy lifestyles occurs too late to prevent childhood obesity and establish lifelong healthy body weights. To break the spiralling cycle of generations of unhealthy body weights in Canadian children, and to reduce the risk of future obesity-related health problems, it is imperative to prevent excessive pregnancy weight gain, GDM and to promote a healthy prenatal and early postnatal lifestyle.

Reversing the obesity epidemic will involve a lifetime of effort by the medical and research communities, however, over the next 3 years, we believe that we may contribute to the solution by using a two-pronged approach by first targeting pregnant overweight and obese women with a healthy lifestyle approach called the Nutrition & Exercise Lifestyle Intervention Program (NELIP) combined with a Family-based Behavioural Treatment (FBBT) that will prevent excessive weight gain and GDM, and promote a healthy fetal environment. The second prong will use this healthy lifestyle (NELIP+FBBT) approach starting at 2 months postpartum continuing to the first year, to minimize postpartum weight retention, encourage breastfeeding, and promote a healthy family lifestyle.

Primary objectives are:

1. To prevent excessive pregnancy weight gain and GDM in order to decrease the incidence of macrosomia and large for gestational age babies
2. To prevent weight retention postpartum and encourage healthy infant feeding practices in order to decrease the risk of developing obesity during the first year of life.

Secondary objectives are:

1. To track pregnancy weight gain and postpartum weight loss, gradually reducing body weight as needed (0.5 kg per week) to achieve and maintain a healthy body weight in the mother
2. To track birth weight and infant growth within the first year of life (at 2, 6 and 12 months), including body weight, height, BMI, and body fatness, using the World Health Organization growth charts as a standard.

Currently, the R. Samuel McLaughlin Foundation-Exercise and Pregnancy Lab at the University of Western Ontario is the only research laboratory in North America actively investigating metabolic changes in exercising pregnant and postpartum women. Our longitudinal aim is to reduce obesity, and chronic disease risks (such as diabetes) in the offspring of overweight and obese women using our two-pronged intervention program, which includes healthy food choices and increased physical activity (NELIP and FBBT) initiated during pregnancy and reinforced in the early postpartum period. With our NELIP team as a cornerstone, and our pilot data already collected, we foresee an opportunity over the next 3 years to contribute to intervention strategies and patient care with emphasis on disease prevention and healthy family lifestyle initiation early in life to reverse the trend of childhood obesity. With a solid research-based initiative from the lab to the community by knowledge translation to health care providers, future health care costs can be reduced by putting prevention-based programs into practice.

ELIGIBILITY:
Inclusion Criteria:

* medically pre-screened for contraindications to exercise
* prior to 16 weeks gestation (pregnancy program)
* singleton pregnancy and pre-pregnancy BMI equal or greater than 25
* before 2 months post delivery (postpartum program)
* BMI equal or greater than 25 (postpartum program)

Exclusion Criteria:

* diagnosed with gestational diabetes or type 2 diabetes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To prevent excessive pregnancy weight gain and GDM to decrease incidence of macrosomia | weekly weight gain during pregnancy and birth
  To prevent excessive pregnancy weight gain on NELIP and GDM in order to decrease the incidence of macrosomia and large for gestational age babies (> 4.0 kg)

SECONDARY OUTCOMES:
To prevent weight retention in the mother and encourage healthy infant feeding practices | 2, 6 and 12 months post delivery
  To prevent weight retention postpartum (gradually reducing body weight as needed by 0.5 kg per week) to achieve and maintain a healthy body weight in the mother and to encourage healthy infant feeding practices in order to decrease the risk of obesity during the first year of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F Mottola, PhD, Principal Investigator — Western University, Canada
Locations (1):
- Exercise and Pregnancy Lab, 2245, 3-M Centre - University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Result] Mottola MF, Giroux I, Gratton R, Hammond JA, Hanley A, Harris S, McManus R, Davenport MH, Sopper MM. Nutrition and exercise prevent excess weight gain in overweight pregnant women. Med Sci Sports Exerc. 2010 Feb;42(2):265-72. doi: 10.1249/MSS.0b013e3181b5419a. PMID 20083959
- [Derived] Hubbard ME, Ruchat SM, Davenport MH, Prapavessis H, Gratton R, McManus R, Giroux I, Hanley AJ, Mottola MF. Impact of an Antenatal Family-based Behavioral Treatment with a Nutrition and Exercise Lifestyle Intervention Program on Infant Weight-for-length at Birth. Int J Behav Med. 2025 Jan 6. doi: 10.1007/s12529-024-10345-8. Online ahead of print. PMID 39762494
- See also: Click for more information about this study. — http://www.uwo.ca/fhs/EPL